CLINICAL TRIAL: NCT05435222
Title: Evaluation of a Male-specific Psychotherapeutic Program for Major Depressive Disorders Compared to Standard Cognitive Behavioral Therapy: a Randomized Controlled Superiority Trial
Brief Title: Evaluation of a Male-specific Psychotherapeutic Program for Major Depressive Disorders
Acronym: MSPP-MDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Walther (Other)
Responsible Party: Sponsor-Investigator, Andreas Walther, Dr. phil., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 000-000-001
Record Dates: First submitted 2020-09-14; First posted 2022-06-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: six-arm randomized controlled superiority trial 2x3 factorial study design Additionally, a healthy control group will be examined, which will undergo only baseline assessments.
  The study is a six-arm randomized controlled superiority trial. Participants will be stratified by testosterone status (eugonadal / hypogonadal) and then randomized into one of the three groups (MSPP, CBT or Waitlist). The study presents a 2x3 factorial study design. In addition, a separate healthy control group will be examined, which will undergo only baseline assessments.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- male-specific psychotherapeutic program (MSPP) (Experimental): In this treatment group, eugonadal depressed men will receive the male-specific adjusted psychotherapy for depressive disorders (MSPP) based on cognitive behavioral principles in a single setting.
  Interventions: Behavioral: Male-specific psychotherapeutic program (MSPP)
- cognitive behavioral therapy (CBT) (Active Comparator): In this treatment group, depressed men will receive standard cognitive behavioral psychotherapy for depressive disorders (CBT) in a single setting.
  Interventions: Behavioral: Cognitive beahvioral therapy (CBT)
- Waitlist (No Intervention): The participants in the Waitlist group are required to complete a waiting period of 36 weeks prior receiving the MSPP.
  As an additional safety measure, participants will be monitored by means of three appointments at week 6, 10 and 14 with a study psychologist. Subsequently, monthly telephone calls at week 18, 22, 26, and 30 are conducted. During these appointments no intervention will occur, while a treatment relationship is to be established so that the patient can describe his specific life circumstances and report possible symptom exacerbations or suicidality.
- male-specific psychotherapeutic program (MSPP) + testosterone treatment (TT) (Experimental): In this treatment group, hypogonadal depressed men will receive the male-specific adjusted psychotherapy for depressive disorders (MSPP) based on cognitive behavioral principles in a single setting. Further participants receive a standard testosterone replacement therapy consisting of testosterone undecanoate administered via deep intramuscular injection.
  Interventions: Behavioral: Male-specific psychotherapeutic program (MSPP)
- cognitive behavioral therapy (CBT) + testosterone treatment (TT) (Active Comparator): In this treatment group, hypogonadal depressed men (blood testosterone ≤ 12.1 nmol/l) will receive standard cognitive behavioral psychotherapy for depressive disorders (CBT) in a single setting. Further participants receive a standard testosterone replacement therapy consisting of testosterone undecanoate administered via deep intramuscular injection.
  Interventions: Behavioral: Cognitive beahvioral therapy (CBT)
- Waitlist + testosterone treatment (TT) (No Intervention): The participants in the Waitlist group are required to complete a waiting period of 36 weeks prior receiving the MSPP. As an additional safety measure, participants will be monitored by means of three appointments at week 6, 10 and 14 with a study psychologist. Subsequently, monthly telephone calls at week 18, 22, 26, and 30 are conducted. During these appointments no intervention will occur, while a treatment relationship is to be established so that the patient can describe his specific life circumstances and report possible symptom exacerbations or suicidality.
  Further participants receive a standard testosterone replacement therapy consisting of testosterone undecanoate administered via deep intramuscular injection.

INTERVENTIONS:
Behavioral: Male-specific psychotherapeutic program (MSPP) — The MSPP for MDD is designed to be used for the acute treatment of depression in men in 18 sessions over a period of 18 weeks. Therapy is delivered weekly with homework bridging every session. Central CBT elements (e.g. behavioral activation, cognitive restructuring) will be retained in MSPP. During implementation of typical CBT techniques, masculine role norms will be considered. One underlying topic will be the potential of multiple masculinities to coexist, being fluid and relational within one man, emphasizing positive aspects of masculinities compatible with psychotherapy for MDD.
  Arms: male-specific psychotherapeutic program (MSPP); male-specific psychotherapeutic program (MSPP) + testosterone treatment (TT)
Behavioral: Cognitive beahvioral therapy (CBT) — This intervention consists of 18 sessions of manualized, standard cognitive behavioral therapy for major depression. Therapy is delivered weekly with homework bridging every session.
  Arms: cognitive behavioral therapy (CBT); cognitive behavioral therapy (CBT) + testosterone treatment (TT)

SUMMARY:
This project aims to evaluate a male-specific psychotherapeutic program (MSPP) for MDD based on cognitive behavioral therapy (CBT). The primary goal is to test the superiority of the MSPP. This will be conducted in two groups of depressed men, namely eudonadal depressed men and hypogonadal depressed men receiving testosterone treatment (TT). In a randomized study design, the MSPP will be compared to a standard CBT and a waitlist control group, resulting in a total of six study groups. Both standardized psychotherapy programs will encompass 18 sessions delivered in a weekly manner, starting at study week 6 and continuing until study week 24. Aligned with the TT-related medical visits of the hypogonadal men, all participants will be followed up with clinical assessments and biosampling at weeks 0, 6, 15, 24, 36. In addition, a separate healthy control group will be examined, which will undergo only baseline assessments.

DETAILED DESCRIPTION:
Background: Although women are twice as likely to suffer from major depressive disorder (MDD) than men, there are still over 100 million men affected by this condition worldwide. Unfortunately, men suffering from MDD seek mental health services about 30% less than women, leaving a large portion of men with unresolved mental health needs. This is reflected in 2-fold higher rates of alcohol use disorder and 4-fold higher rates of completed suicide amongst men, while MDD is considered a prime risk factor for both. A case is made for male-typical MDD phenotypes with differing symptom presentation often unrecognized by clinicians. Although cognitive behavioral therapy (CBT) represents an effective treatment for MDD, conformity to traditional masculinity norms based on stoicism, self-reliance, and restrictive emotionality often hinder men from engaging in psychotherapy. Therefore, a need to address this diagnostic and treatment gap emerges, while recent studies have identified a lack of male-specific psychotherapeutic programs (MSPP) that could persuade more men to take on psychotherapy based on a male-tailored nature, focusing on male-specific topics and being introduced in male-typical environments.

Method and study procedures: In total, 144 depressed men aged between 25 and 50 will be recruited. After Screening procedures, included participants are stratified by testosterone status (hypogoadal vs. eugonadal) and randomized to one of the conditions: MSPP, CBT, Waitlist. This results in six intervention groups (MSPP, CBT, Waitlist, MSPP+TT, CBT+TT, Waitlist+TT). Hypogonadal men will receive testosterone treatment administered at the Andrology-Urology Center (Uroviva). MSPP and CBT intervention groups will receive weekly therapy sessions for MDD over 18 weeks. All participants will be invited to a total of five examination appointments (weeks 0, 6, 15, 24, 36) at the psychological institute of the university of Zurich. In addition, a separate healthy control group will be examined, which will undergo only baseline assessments.

Expected results: Compared to the waitlist control groups, the treatment groups are expected to be more effective and efficacious (depression score reduction of ≥50%) at week 24 and at follow-up week 36. The MSPP, compared to CBT, is expected to show higher effectiveness and efficacy for depression symptoms, higher acceptability and a greater reduction of gender role conflict. In addition, it is expected that the initially hypogonadal men will have increased symptom improvement due to TT as compared to the eugonadal men in the parallel groups and that TT receiving men show an adjunct effect of added psychotherapy as compared to men in the waitlist.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex
2. Age between 25 - 50 years
3. German speaking
4. Current major depression (assessed by SCID-5)
5. Informed consent as documented by signature

Exclusion Criteria:

1. Inability to give informed consent
2. Prior hormonal (testosterone) treatment
3. Prior mental health disorder
4. Current or previous psychopharmacological treatment
5. Current or previous psychological treatment for any psychological disorder

   - Exception for persistent depressive disorder (Dysthymia) and alcohol/substance use disorder of mild degree (SCID-5, 1 - 3 criteria met)
6. Comorbidities of major depression with any other psychological disorder
7. Severe physical disorder that requires priority treatment
8. Any of the following physical conditions, particularly relevant in regard to testosterone treatment:

   * Diagnosed prostate cancer
   * Prostatic intraepithelial neoplasia (PIN)
   * Severe lower urinary tract symptoms
   * Erythrocytosis Sleep apnea, diagnosed but untreated
9. Current treatment with:

   * Thyroid hormones
   * Finasteride
   * Antiepileptic drugs
   * Anabolic compounds
   * Hypnotic medication more than 2 nights/week for the treatment of insomnia
   * Long-acting benzodiazepines
   * Antipsychotic medication
   * Drugs that affect serum testosterone
10. Genetic / hormonal disorders:

    * Klinefelter's syndrome
    * Cushing's disease
    * Addison's disease
    * Hashimoto Thyroiditis

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline observer assessed depressive symptomatology to post treatment | baseline / 24 weeks
  Observer assessed depressive symptomatology measured with the Hamilton Depression Rating Scale (HDRS-21)
Changes in the clinical symptomatology from baseline to post treatment | baseline / 24 weeks
  Observer assessed clinical symptomatology measured with the Clinical Global impression Scale (CGI-S/I)
Change from baseline male typical depressive symptomatology to post treatment | baseline / 24 weeks
  Self-reported male typical depression symptoms including externalizing behavior such as aggression, risk taking, or alcohol consumption measured with the Male Depression Risk Scale (MDRS-22)
Change from baseline self-reported depressive symptomatology to post treatment | baseline / 24 weeks
  self-reported depressive symptomatology measured with the Beck Depression Inventory (BDI-II)
Changes in gender role conflict | baseline / 24 weeks
  Self-reported symptoms of gender role conflict measured with the Gender Role Conflict Scale (GRCS-16)
Drop out | at follow up week 36
  Acceptability: Proportion of men who withdraw for any reason (dropout) will be recorded and if dropped out participants consent, a dropout interview will be conducted to examine the reasons for dropout.
Achieved remission | post treatment week 24
  Proportion of participants, that achieved depressive symptom remission (assessed by structured clinical interview [SCID-5-CV] for DSM-V disorders)
Changes in the therapeutic alliance quality | week 6 / week 24
  Self reported working alliance quality with the therapist

SECONDARY OUTCOMES:
Skala Suizidales Erleben und Verhalten (SSEV-9) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported suicidal experience and behavior
Suicide Cognitions Scales (SCS-18) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported attitudes toward suicide
Problematic Pornography Consumption Scale (PPCS-18) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported pornography use and problematic consumption
Alcohol Use Disorder Test 10 (AUDIT-10) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported alcohol consumption symptomatology
International Index of Erectile Function 15 (IIEF-15) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported sexual dysfunction and libido symptomatology
Perceived Stress Scale (PSS-10) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported subjective stress
Generalized Anxiety Disorder (GAD-7) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported general anxiety
Conformity Masculine Norms Inventory (CMNI-30) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported conformity to traditional male role norms
Male Role Norms Inventory - Short Form (MRNI-SF-21) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported socially learned male role norms
Precarious Manhood Beliefs Scale (PMB-4) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported precarious manhood beliefs
Loneliness Scale (LS-20) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported feeling of loneliness and social isolation
Self-Compassion Scale D (SCS-D 10) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported Positive attitude towards oneself in difficult life situations
Emotion Regulation Questionnaire (ERQ-10) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported tendency to re-evaluate / suppress emotions
General Belongingness Scale (GBS) | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Self-reported achieved belongingness
CIDI-Traumaliste (CIDI-T-12) | baseline / week 6 / post treatment week 24 / follow up week 36
  Assessment of self-reported traumatic experiences over the life span
International Trauma Questionnaire (ITQ-18) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported core symptoms of post-traumatic stress disorder and complex post-traumatic stress disorder
Agression Questionnaire Buss and Perry (AQ-BP) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported anger and aggression symptomatology
Fragebogens zum Körperbild (FKB-6) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported attitudes towards one's own and an ideal body image
Male Body Attitudes Scale-Revised (MBAS-R-15) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported male-specific body (dis)satisfaction
Body Appreciation Scale 2 (BAS-2-10) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported assessment of a positive body image
Stigma questionnaire (STIG-9) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported experienced stigma for suffering from a mental illness
Self-stigma of seeking psychological help (SSOSH-10) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported experienced stigma of seeking help
SHAME Questionnaire (SHAME-21) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported physical, cognitive and existential shame
Test of Self-Conscious Affect (TOSCA-16) | baseline / week 6 / post treatment week 24 / follow up week 36
  Assessment of susceptibility to guilt, shame, externalization, and unconcern (self-report questionnaire).
Toronto Alexithymia Scale (TAS-20) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported difficulty identifying and describing emotions
Multidimensional Self-Concept Scale (MSCS) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported self-concept (self-worth)
Arnett Inventory of Sensation Seeking (AISS-20) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported seeking of intense experiences including risky behavior
Need to Belong Scale (NTBS-10) | baseline / week 6 / post treatment week 24 / follow up week 36
  Self-reported motivation to be accepted by others and avoidance of rejection by others

OTHER OUTCOMES:
Body composition | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Body composition is determined by using bioelectrical impedance analysis (BIA)
Blood testosteron | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Blood samples are collected at each study visit to assess blood testosterone
Hair testosterone | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Hair samples are collected at each study visit to assess hair testosterone
Grip strength | baseline / week 6 / week 15 / post treatment week 24 / follow up week 36
  Grip strength will be assessed with a basic hydraulic hand dynamometer at each study visit

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Walther, PhD, Principal Investigator — University of Zurich
Locations (1):
- Ambulatory for Cognitive Behavioral Therapy and Behavioral Medicine of the University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walther A, Ehlert U, Schneeberger M, Eggenberger L, Fluckiger C, Komlenac N, Heald A, Rice T, Palm S, Seidler ZE, Ogrodniczuk JS, Oliffe JL, Rice SM, Kealy D, Weber R, Zimmermann D. Evaluation of a male-specific psychotherapeutic program for major depressive disorder compared to cognitive behavioral therapy and waitlist: study protocol for a six-arm randomized clinical superiority trial examining depressed eugonadal and hypogonadal men receiving testosterone. Front Psychiatry. 2023 Jun 21;14:1129386. doi: 10.3389/fpsyt.2023.1129386. eCollection 2023. PMID 37415687